CLINICAL TRIAL: NCT05021692
Title: Efficiency of the Web-Based Support Program Based on the Health Promotion Model in Pregnant Women With Preeclampsia
Acronym: preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Büşra Yılmaz, Msc, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: busrayılmaz
Record Dates: First submitted 2021-07-10; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Healthy Lifestyle; Preeclampsia; Pregnancy; Renal Disease
Keywords: healthy life; web-based support; risky pregnancy; preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, single-blind, randomized-controlled type experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group: Pregnant women with preeclampsia who receive a web-based support program based on the Health Promotion Model in addition to routine clinical care will form the intervention group.
  Interventions: Behavioral: Web-based support program for pregnant women with preeclampsia based on the Health Promotion Model
- Control (No Intervention): Pregnant women who receive routine clinical care applied to pregnant women with preeclampsia will constitute the control group.

INTERVENTIONS:
Behavioral: Web-based support program for pregnant women with preeclampsia based on the Health Promotion Model — support program
  Other Names: Routine clinical care applied to pregnant women with preeclampsia
  Arms: Intervention

SUMMARY:
In the literature, it has been reported that health promotion model-based care approaches are beneficial in gaining positive healthy lifestyle behaviors, taking responsibility for the individual's health and increasing the quality of life. It is thought that the health promotion model in pregnant women with preeclampsia will positively affect the healthy lifestyle behaviors and self-efficacy level of pregnant women by ensuring active participation of pregnant women in symptom management, reduce the stress of the pregnant and positively affect maternal and fetal-neonatal health outcomes. In line with this information, it was aimed to determine the effect of the web-based support program based on the health promotion model on maternal infant health in pregnant women with preeclampsia.

DETAILED DESCRIPTION:
Research Hypotheses H1a: The web-based support program based on the Health Promotion Model enables the pregnant woman to monitor blood pressure, weight, edema.

H1b: The web-based support program based on the Health Promotion Model increases the baby's postpartum first-minute apgar score, fifth-minute apgar score, and prevents the baby's respiratory distress.

H1c: Web-based support program based on the Health Promotion Model positively affects fetal-neonatal health outcomes.

H1d: The web-based support program based on the Health Promotion Model reduces the stress of pregnant women related to their own and their baby's health.

H1e: The web-based support program based on the Health Promotion Model enables the mother to make decisions about her health and to participate in decisions about her health.

Research Type It is a prospective, single-blind, randomized controlled-type experimental study using a pre-test-post-test layout. Research Place and Time The study is planned to be carried out with pregnant women who applied to Obstetrics and Gynecology clinics in Istanbul University - Cerrahpaşa Cerrahpaşa Medical Faculty Hospital. After the research ethics committee and institution permissions are obtained, it is planned to begin the application phase with patients in June 2021.

Study Population and Sample The universe of the study will be composed of pregnant women who applied to Obstetrics and Gynecology clinics at the dates of the research at Istanbul University - Cerrahpaşa Cerrahpaşa Medical Faculty. In order to calculate the sample size, the power of the study was calculated in the G * Power (v3.1.7) program. The total score of the Healthy Lifestyle Behaviors Scale was used as the main parameter in the study. In the study, the HLBS total score after healthy lifestyle behaviors training was found to be 125.11 ± 16.86 in the control group, and 138.22 ± 27.88 in the intervention group, after training on healthy lifestyle behaviors for women at 20-24 weeks of gestation (1). In the statistical analysis made on the basis of the results of this study, the alpha reliability level of the study was taken as 0.05 and the power was 80%, and the minimum number of pregnant women required for each group was determined as 39 according to the HLBS score in the two-way hypothesis analysis. Considering that there may be losses during the working process, it is planned to include 45 people to each group. As a result, according to the results of the power analysis, the number of pregnant women to be included in the study was 45 for each group as an experimental and a control group, and the total number of pregnant women to be included in the study was 90.

Working Groups:

Intervention group: Pregnant women with preeclampsia who receive a web-based support program based on the Health Promotion Model in addition to routine clinical care will form the intervention group.

Control group: Pregnant women who receive routine clinical care applied to pregnant women with preeclampsia will constitute the control group.

C.1.2.1. Facts

Inclusion Criteria:

Having been diagnosed with preeclampsia

* Having internet access
* Being older than the 20th gestational week
* Over the age of 18
* Having a single live fetus
* No diagnosed psychiatric disease
* Being literate
* Being willing to participate in the study.

Exclusion Criteria from the Study:

* Not having internet access or not knowing how to use it
* Having an accompanying chronic disease
* Inability to communicate in Turkish
* Having inpatient treatment at the hospital C.1.2.2. Methods to be Used in the Study The study is planned to be carried out with 90 pregnant women diagnosed with preeclampsia who applied to Obstetrics clinics or received treatment at Istanbul University - Cerrahpaşa Cerrahpaşa Medical Faculty at the time of the research.

Before working with pregnant women, a web site will be created and opinions of 10 experts will be taken on the suitability of the site. The web page expert opinion form will be carried out under the guidance of the DISCERN Guidelines (Appendix 1), and the consistency between the scores of the experts will be evaluated with the Kendall Conformity Coefficient. Information on the features of the website is given in Annex 2. After the expert opinions, the website will be finalized and the pre-application of the study will be made. A pre-application will be done with 10% of the participants (n = 5) of the initiative group, and these participants will not be included in the results of the study. Pregnant women who meet the inclusion criteria will be randomly distributed to the intervention and control groups through a randomized procedure. For randomization in this distribution, randomization was performed using a computer program module used in controlled studies (http://www.randomizer.org/form.htm). Pregnant women to be included in the study according to the order of the researcher meeting the pregnant in the hospital; to the initiative group; (7, 41, 39, 69, 79, 49, 12, 14, 72, 15, 13, 59, 60, 63, 73, 22, 67, 68, 42, 56, 77, 54, 66, 33, 30 5, 25, 32, 26, 86, 81, 18, 20, 55, 11, 62, 29, 85, 84, 45, 40, 28, 47, 17, 35) to the control group; (71, 37, 54, 23, 84, 18, 53, 29, 40, 68, 44, 72, 75, 32, 11, 39, 48, 16, 30, 59, 87, 6, 20, 2, 66 , 33, 62, 10, 35, 74, 4, 56, 90, 63, 14, 12, 21, 89, 25, 9, 67, 57, 69, 38, 81) placed by matching Until the data reaches the sample size, the experimental and control groups will be collected together. The study will be added to the protocol registration system where interventional research is recorded (clinicaltrials.gov) and the NCT number will be obtained for the study.

In the first interview with pregnant women, an explanation about the study will be made, and the consent of the participants will be obtained through the informed consent form (Annex 3, Annex 4) prepared separately for the intervention and control group. In both groups, at the first interview, "Participant introduction form (Appendix 5)", "Healthy Lifestyle Behaviors Scale (HLBS) (Appendix 6)", "Prenatal Distress Scale (PBI)" (Appendix 7) "and" Self-efficacy Scale (AAS) ) (Annex 8) "will be applied. Both groups will be given a brochure about preeclampsia at the first encounter. The web site will be introduced to the initiative group, a username and password will be given to login, and how to use the web site will be taught. If pregnant women do not log in to the site within five days after the password is given, a reminder will be made via e-mail or telephone. If they still do not log in to the site in case of a reminder, they will be disabled. The planned training program will be started with the first entry of pregnant women to the website. It will be ensured that pregnant women complete the six modules with the following topics in two weeks. After each module, 5-6 questions will be added, if the participant answers the questions correctly, they will be able to switch to the next module. The researcher will track the completion status of the modules over the course of two weeks. Pregnant women will be able to complete the modules 24 hours a day whenever they are available.

Module titles:

* What is preeclampsia and what are the danger signs in preeclampsia?
* How can preeclampsia symptoms be followed at home?
* What can a pregnant woman do to adapt to the treatment of preeclampsia?
* What should be done to improve health in preeclampsia?
* How should a pregnant with preeclampsia monitor herself in the postpartum period?
* What should a pregnant woman with preeclampsia do for the risk of developing preeclampsia in the next pregnancy? Participants will evaluate the usefulness / satisfaction of the training through the Vizuel Analog Scale after each module. Web-based support program subjects, content and training plan, "Topic and content plan, module purpose, learning objectives, training period and training materials" and "Web-based support program based on health development model" are given in Annex 9. No intervention will be made to the control group, and the control group will receive routine care according to the hospital protocol. Two weeks after the first interview, "HLBS", "AAS", "PBL" and "Self-monitoring form of the pregnant woman (Appendix 10) will be applied to both groups twice with two-week intervals.

Postpartum monitoring will be performed on postpartum 0, 1, and 2 days using the "Postpartum evaluation form (Appendix 11)". Data collection tools will be sent to the control group via e-mail, the participants will be called from time to time and the status of filling out the forms will be questioned. The initiative group will fill out the questionnaires on the website and will be called by the researcher at least once a week. Pregnant women will be able to conduct investigative interviews on the meet with experts platform (Google meet, zoom, etc.) when they need it. The initiative group will be able to chat with other participants from the forum page on the website. When necessary, they will be able to communicate with the researcher both on the website and on the phone. A "Frequently Asked Questions" section will be created by the researcher on the website, and the participants in the initiative group will be able to benefit from that section whenever they want. Postpartum 2nd day, the initiative group will evaluate the usability of the website with the "System Usability Scale (Annex 12)". Process evaluation form will be used in the study. Process evaluation is used to document and monitor the implementation of the program. A process evaluation plan will be implemented in each of the stages of the planning, method, data collection tools, implementation and evaluation of the study. In the first interview with pregnant women, an explanation about the study will be made, and the consent of the participants will be obtained through the informed consent form prepared separately for the intervention and control group. "Participant introduction form", "Healthy Lifestyle Behaviors Scale", "Prenatal Distress Scale" and "Self-efficacy Scale" will be applied to both groups in the first interview. Both groups will be given a brochure about preeclampsia at the first encounter. The web site will be introduced to the initiative group, a username and password will be given to login, and how to use the web site will be taught. If pregnant women do not log in to the site within five days after the password is given, a reminder will be made via e-mail or telephone. If they still do not log in to the site in case of a reminder, they will be disabled. The planned training program will be started with the first entry of pregnant women to the website. It will be ensured that pregnant women complete the six modules with the following topics in two weeks. After each module, 5-6 questions will be added, if the participant answers the questions correctly, they will be able to switch to the next module. The researcher will track the completion status of the modules over the course of two weeks. Pregnant women will be able to complete the modules 24 hours a day whenever they are available.

Module titles:

* What is preeclampsia and what are the danger signs in preeclampsia?
* How can preeclampsia symptoms be followed at home?
* What can a pregnant woman do to adapt to the treatment of preeclampsia?
* What should be done to improve health in preeclampsia?
* How should a pregnant with preeclampsia monitor herself in the postpartum period?
* What should a pregnant woman with preeclampsia do for the risk of developing preeclampsia in the next pregnancy? Participants will evaluate the usefulness / satisfaction of the training through the Vizuel Analog Scale after each module. No intervention will be made to the control group, and the control group will receive routine care according to the hospital protocol. Two weeks after the first interview, "Healthy lifestyle behaviors scale", "Self-efficacy scale", "Prenatal distress scale" and "Pregnant's self-monitoring form will be applied to both groups two weeks apart.

Postpartum monitoring will be carried out on postpartum 0, 1, and 2 days using the "Postpartum evaluation form". Data collection tools will be sent to the control group via e-mail, the participants will be called from time to time and the status of filling out the forms will be questioned. The initiative group will fill out the questionnaires on the website and will be called by the researcher at least once a week. Pregnant women will be able to conduct investigative interviews on the meet with experts platform (Google meet, zoom, etc.) when they need it. The initiative group will be able to chat with other participants from the forum page on the website. When necessary, they will be able to communicate with the researcher both on the website and on the phone. A "Frequently Asked Questions" section will be created by the researcher on the website, and the participants in the initiative group will be able to benefit from that section whenever they want. On the 2nd day of postpartum, the initiative group will evaluate the usability of the website with the "System Usability Scale". Process evaluation form will be used in the study. Process evaluation is used to document and monitor the implementation of the program. A process evaluation plan will be implemented in each of the stages of the planning, method, data collection tools, implementation and evaluation of the study. At every stage of the study, it was prepared in accordance with the parameters of fidelity, dose delivered, dose received, reach, recruitment and content / context (contex) parameters.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with preeclampsia
* Having internet access
* Being older than the 20th gestational week
* Over the age of 18
* Having a single live fetus
* No diagnosed psychiatric disease
* Being literate
* Being willing to participate in the study.

Exclusion Criteria:

* Not having internet access or not knowing how to use it
* Having an accompanying chronic disease
* Inability to communicate in Turkish
* Having inpatient treatment at the hospital

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Web-based support program based on the Health Promotion Model positively affects fetal-neonatal health outcomes. | 6-12 months
  The mother feels at least 10 movements in two hours in the follow-up of the baby movements.
  Postpartum first and fifth minute Apgar score is seven or more out of 10 points.
  The newborn did not need intensive care support. The newborn had no respiratory distress.
The web-based support program based on the Health Promotion Model reduces the stress of pregnant women regarding their own and their baby's health. | 6-12 months
  There was a decrease in the scores of the pregnant women in the intervention group from the Prenatal Distress Scale, and the pregnant women in the intervention group had a statistically lower score on the Prenatal Distress Scale than the pregnant women in the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Büşra Yılmaz, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Asci O, Rathfisch G. Effect of lifestyle interventions of pregnant women on their dietary habits, lifestyle behaviors, and weight gain: a randomized controlled trial. J Health Popul Nutr. 2016 Feb 24;35:7. doi: 10.1186/s41043-016-0044-2. PMID 26911204